CLINICAL TRIAL: NCT04893551
Title: Phase 1b, Multicentre, Multiple Ascending Dose, Safety, Pharmacokinetic, and Pharmacodynamic Study of Tilvestamab (BGB149) in Relapsed, Platinum-resistant, High-grade Serous Ovarian Cancer (HGSOC) Patients
Brief Title: A Study of Tilvestamab (BGB149) in Relapsed, Platinum-resistant, High-grade Serous Ovarian Cancer (HGSOC) Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: After completion of all planned dose levels in the dose escalation phase, the sponsor decision was not to continue with expanding the cohorts of any of the dose levels, using the existing study design.
Sponsor: BerGenBio ASA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB149-102; 2020-001382-36 (EudraCT Number)
Record Dates: First submitted 2021-05-17; First posted 2021-05-19 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tilvestamab (Experimental): Participants will receive tilvestamab at a low starting dose level (Cohort A) given via intravenous (IV) infusion every 2 weeks. Dose escalations to subsequent cohorts (Cohort B and Cohort C) will be decided by the Protocol Steering Committee (PSC) after review of all Cycle 1 (28 days cycle) safety and pharmacokinetics (PK) data up to Cycle 1 Day 22 for all participants in the ongoing cohort.
  Interventions: Biological: Tilvestamab

INTERVENTIONS:
Biological: Tilvestamab — Tilvestamab will be administered as IV infusion.
  Other Names: BGB149

SUMMARY:
The primary purpose is to assess the safety and tolerability of tilvestamab following IV administration of multiple doses to participants with HGSOC who have been treated with at least 1 complete course of platinum-based chemotherapy and whose disease has relapsed with platinum resistance ([PRR]-HGSOC) and to determine the plasma pharmacokinetics (PK) exposure by comprehensive profiling (at single dose and steady-state) of multiple ascending doses of tilvestamab.

ELIGIBILITY:
Inclusion Criteria:

* Females of non-childbearing potential at the time of provision of informed consent
* Ability to understand and provide written confirmation of informed consent after reading study information, discussion with the investigator, and adequate time to decide on participation
* Consents to storage of study-related samples and data for exploratory use
* Histologically confirmed HGSOC
* Platinum-resistant relapsed disease; defined as progressive disease based on imaging within <= 6 months from completion of most recent regimen

Exclusion Criteria:

* Primary platinum-refractory disease (ie, progression during the first platinum regimen or within 4 weeks of completion of the first platinum regimen) with rapid progression and life-threatening disease manifestation
* Life expectancy < 6 months
* Concurrent anticancer therapy
* Participants who are breastfeeding
* Known uncontrolled central nervous system metastases. Participants without known brain metastases do not require radiological imaging prior to enrolment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse events (AEs) and Serious AEs (SAEs) | Up to 2.5 years
  An AE is any symptom, physical sign, syndrome, or disease that either emerges during the study or, if present at Screening, worsens during the study, regardless of the suspected cause of the event. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Number of Participants with Laboratory Abnormalities | Up to 2.5 years
  Number of participants with laboratory (haematology, coagulation, clinical chemistry, serum inflammatory cytokine profile, and urinalysis) abnormalities will be reported.
Number of Participants with Vital Sign Abnormalities | Up to 2.5 years
  Number of participants with vital sign (supine blood pressure [BP], heart rate, oral temperature, and respiratory rate) abnormalities will be reported.
Number of Participants with Electrocardiogram (ECG) Abnormalities | Up to 2.5 years
  Number of participants with resting triplicate 12-lead ECG abnormalities will be reported.
Number of Participants with Physical Examinations Abnormalities | Up to 2.5 years
  Number of participants with physical examinations abnormalities will be reported.
Number of Participants with Concomitant Medication Use | Up to 2.5 years
  Number of participants with concomitant medication use will be reported.
Maximum Concentration (Cmax) | Up to 140 days
  Cmax will be determined directly from the concentration-time profile.
Time to Cmax (Tmax) | Up to 140 days
  Time to Cmax will be determined directly from the concentration-time profile.
Area Under the Concentration-time Curve (AUC) From Predose (Time 0) to the end of the Dosing Period (AUC0-tau) | Up to 140 days
  AUC0-tau will be calculated using the linear-log trapezoidal rule.
AUC From Predose (Time 0) to the Time of the Last Quantifiable Concentration (AUClast) | Up to 140 days
  AUClast will be calculated using the linear-log trapezoidal rule.
AUC From Predose (Time 0) to 168 Hours Postdose (AUC0-168 ) | Predose up to 168 hours postdose
  AUC0-168 is AUC from predose (time 0) to 168 hours postdose.
Terminal Elimination Rate Constant (Lambda[z]) | Up to 140 days
  Lambda[z] will be determined by selection of at least 3 data points on the terminal phase of the concentration-time curve.
Terminal Elimination Half-life | Up to 140 days
  Terminal elimination half-life calculated as: ln2/Lambda[z]
Total body clearance (CL) | Up to 140 days
  CL is defined as total body clearance.

SECONDARY OUTCOMES:
Number of Participants with Anti-drug Antibodies (ADAs) | Up to 2.5 years
  Number of participants with ADAs will be reported.
Number of Participants with Neutralizing Antibodies (NAbs) | Up to 2.5 years
  Number of participants with NAbs will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Akil Jackson, Study Director — BerGenBio ASA
Locations (9):
- Haukeland University Hospital Bergen, Bergen, Norway
- National University Hospital, Singapore, Singapore
- South Korea (3):
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System- Severance Hospital, Seoul
- United Kingdom (4):
  - Western General Hospital, Edinburgh
  - Guys and St Thomas' NHS Foundation Trust, London
  - Imperial College London, Hammersmith Hospital, London
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification [text, tables, figures and appendices].
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Proposal should be directed to HYPERLINK "mailto:clinical@bergenbio.com" clinical@bergenbio.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Sooi K, Tan TZ, Kim JW, Lee JY, Kim BG, Micklem D, Jackson A, Pinato DJ, Gourley C, Kristeleit R, Blagden SP, Bjorge L, Tan DSP. A phase 1b, multicentre, dose escalation, safety and pharmacokinetics study of tilvestamab (BGB149) in relapsed, platinum-resistant, high-grade serous ovarian cancer (PROC) patients. Br J Cancer. 2025 Oct;133(6):896-908. doi: 10.1038/s41416-025-03090-6. Epub 2025 Jul 22. PMID 40696160